CLINICAL TRIAL: NCT00240812
Title: A Comparative Study of Coadministered Doses of Ibuprofen and Pseudoephedrine HCl and Each Drug Alone in the Treatment of Primary Nocturnal Enuresis in Children
Brief Title: A Study to Determine if Ibuprofen in Combination With Pseudoephedrine HCl is More Effective Than Each Drug Alone in the Treatment of Nighttime Bedwetting
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johnson & Johnson Consumer and Personal Products Worldwide (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR002497
Record Dates: First submitted 2005-10-14; First posted 2005-10-18 (Estimated); Last update posted 2011-06-29 (Estimated); Status verified 2011-06

CONDITIONS: Enuresis
Keywords: nocturnal enuresis; bedwetting; ibuprofen
MeSH Terms: conditions — Enuresis; Nocturnal Enuresis | interventions — Ibuprofen; Pseudoephedrine

INTERVENTIONS:
Drug: ibuprofen; pseudoephedrine HCl

SUMMARY:
The purpose of the study is to determine if ibuprofen in combination with pseudoephedrine HCl in the treatment of nightime bedwetting in children is more effective than each drug alone and if the individual drugs are more effective than placebo.

DETAILED DESCRIPTION:
The objective of this double-blind, placebo-controlled, randomized, parallel-group study is to determine whether the effectiveness of ibuprofen in combination with pseudoephedrine HCl is greater than the individual drugs alone and greater than placebo for the treatment of nighttime bedwetting in children. After a screening visit, parents of eligible patients are to record in a diary, the number of urinations and wet and dry nights. Patients then return and those who continue to be eligible are randomized to study medication, which they will take for two weeks. Patients are randomized into four treatment groups, and the dose of treatment medication is determined based on body weight. The four treatment groups are: 12.5 mg of ibuprofen suspension/kg of body weight (200-450 mg of ibuprofen) plus 15 mg or 30 mg of pseudoephedrine HCl, 12.5 mg of ibuprofen suspension / kg of body weight (200 - 450 mg of ibuprofen) plus placebo suspension, or two doses of placebo suspension. The primary efficacy measurement is the mean reduction in wet nights, for the 14-day baseline period to the 14-day treatment period. Safety assessments consist of monitoring adverse events, physical examination and assessment of vital signs. The study hypothesis is that ibuprofen in combination with pseudoephedrine HCl has a greater effect in the treatment of nighttime bedwetting than either ibuprofen or pseudoephedrine HCl alone, and the combination is well tolerated. Treatment medication are an oral suspension, expressed as mg/kg body weight. Patients will receive 1 of 4 treatments for 2 weeks: ibuprofen (12.5 mg/kg of body weight) plus 15 or 30 mg of pseudoephedrine, ibuprofen (12.5 mg/kg of body weight) + placebo, 15 or 30 mg of pseudoephedrine, or placebo

ELIGIBILITY:
Inclusion Criteria:

* Subject has nighttime bedwetting
* between the 5th and 95th percentiles for weight based on age and gender
* has a minimum of eight wet nights per 14 days of the baseline period
* healthy with no symptoms of any other complicating disease as determined by medical history review, physical examination, and clinical laboratory tests.

Exclusion Criteria:

* Subject has daytime urinary incontinence or abnormal bowel habits (i.e. fecal incontinence or constipation)
* has had episodes of dryness lasting one month or longer, at any time in the past
* has a medical condition which may be relevant to participation in the study
* has a known sensitivity or allergy to the study medications.

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 318 (Actual)
Dates: Study Completion 2002-11 (Actual)

PRIMARY OUTCOMES:
The mean reduction in wet nights from the 14-day baseline period to the 14-day treatment period.

SECONDARY OUTCOMES:
The proportion of subjects with at least a 50% reduction in wet nights from baseline; the mean number of wet nights during the 14 days of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: McNeil Consumer & Specialty Pharmaceuticals, a Division of Mc Neil-PPC, Inc. Clinical Trial, Study Director — McNeil Consumer & Specialty Pharmaceuticals, a Division of McNeil-PPC, Inc.

REFERENCES:
- [Derived] Caldwell PH, Codarini M, Stewart F, Hahn D, Sureshkumar P. Alarm interventions for nocturnal enuresis in children. Cochrane Database Syst Rev. 2020 May 4;5(5):CD002911. doi: 10.1002/14651858.CD002911.pub3. PMID 32364251
- See also: A Study to Determine if Ibuprofen in Combination with Pseudoephedrine HCl is More Effective Than Each Drug Alone in the Treatment of Nighttime Bedwetting — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=905&filename=CR002497_CSR.pdf